CLINICAL TRIAL: NCT02737618
Title: 14-Day Cumulative Irritation Patch Test in Subjects With Normal Skin - Chameleon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ST-7611
Record Dates: First submitted 2016-03-22; First posted 2016-04-14 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Dermal Irritation

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes

ARMS (1):
- Healthy subject (Experimental): Healthy subjects exposed to Trojan "Chameleon" Personal Lubricant applied by occlusive patch
  Interventions: Device: Trojan "Chameleon" Personal Lubricant

INTERVENTIONS:
Device: Trojan "Chameleon" Personal Lubricant — silicone base with sensate

SUMMARY:
to determine the ability of the test article to cause irritation to the skin of humans under controlled patch test conditions

ELIGIBILITY:
Inclusion Criteria:

* male or female, 18-70 years of age, in general good health
* normal skin
* free of any systemic or dermatologic disorder which, in the opinion of the investigative personnel, will interfere with the study results or increase the risk of adverse events
* of any skin type or race providing the skin pigmentation will allow discernment of erythema
* agree to complete a medical history and concomitant medication form
* read, understand and sign informed consent

Exclusion Criteria:

* have any visible skin disease at the study site which, in the opinion of the investigative personnel, will interfere with the evaluation
* are receiving systemic or topical drugs or medication which, in the opinion of the investigative personnel, will interfere with the study results
* have psoriasis and/or active atopic dermatitis/eczema
* have a known sensitivity to cosmetics, skin care test articles, or topical drugs as related to the test article being evaluated
* are females who are pregnant or breastfeeding or become pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Dosik, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research Inc, Fair Lawn, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Subject
Started | 43
Completed | 34
Not Completed | 9
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subject
Number analyzed (Participants) | 34
Age, Customized [Count of Participants; unit: Participants]
  18-69 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Showed Erythema Based on 5 Point Scoring Scale
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subject
Number analyzed (Participants) | 34
Participants | 0

2. Primary Outcome: Number of Subjects That Showed Edema Based on the 5 Point Scoring Scale
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Subject
Number analyzed (Participants) | 34
Participants | 0

ADVERSE EVENTS:
Arm/Group | Healthy Subject
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality agreement in place with PI